# Confidential

# **Statistical Analysis Plan**

## For the Clinical Trial of Protocol BTF16-AP-401

A pilot study to evaluate efficacy and safety of hydrophilic polyurethane foam dressing in patients with pressure ulcer

| Sponsor | Mundipharma Pte Ltd. |
|-----------------------|----------------------|
| Protocol Version/Date | 1.3/19AUG2016 |
| CRF Version/Date | 1.2/19AUG2016 |
| SAP Version/Date | 1.0/27OCT2016 |

**ADM Korea Inc.** 

## Prepared by

| | Hak-Jo Kim | | |
|----------|------------------------------|-----------|--------------------|
| | Name (BS)<br>ADM Korea Inc. | Signature | Date (DD/MMM/YYYY) |
| Reviewed | & Approved by | | |
| | Jong-Eon Lim | | |
| | Name (CRM)<br>ADM Korea Inc. | Signature | Date (DD/MMM/YYYY) |
| | Sung-Hun Park | | |
| | Name (BSM)<br>ADM Korea Inc. | Signature | Date (DD/MMM/YYYY) |
| | Hyun-Jae Kim | | |
| | Name (DSM)<br>ADM Korea Inc. | Signature | Date (DD/MMM/YYYY) |
| | Harsha Arumugam | | |
| | Name<br>Mundipharma Pte Ltd | Signature | Date (DD/MMM/YYYY) |

## - Contents -

| 1. Objective | 5 |
|-------------------------------------------------------------|----|
| 2. Purpose of Study | 5 |
| 3. Study Design | 5 |
| 4. Inclusion/Exclusion Criteria | 6 |
| 5. Discontinuation/Withdrawal and Early Completion Criteria | 7 |
| 6. Statistical Analysis Population | 8 |
| 7. Analysis of Endpoints | 8 |
| 8. Statistical Methodology by Endpoints | 10 |
| 9. Handling Missing Values | 11 |
| 10. Midterm Analysis | 12 |
| 11. Others | 12 |
| 12. Dummy Table List | 13 |
| 13. TLFs | 16 |

#### **Abbreviation**

ADE : Adverse Device Effect

AE : Adverse Event

ALP : ALkaline Phosphatase

ATC : Anatomical Therapeutic Chemical

BS : Biostatistician

BSM : Biostatistician Manager

CRM : Clinical Research Manager

CS Clinically Significant

CSSC : Clinical Signs and Symptoms Checklist

FAS : Full Analysis Set

LOCF : Last Observation Carried Forward

MedDRA : Medical Dictionary for Regulatory Activities

NPUAP : National Pressure Ulcer Advisory Panel

PUSH : Pressure Ulcer Scores for Healing

SADE : Serious Adverse Device Effect

SAE : Serious Adverse Effect

WBC : White Blood Cell

1. Objective

The Statistical Analysis Plan is a guideline for Protocol No.BTF16-AP-401 to minimize the bias and maximize the

precision so that the final results, conclusion, application and the entire details regarding proposed analysis of

the clinical trial can be reliably evaluated.

2. Purpose of Study

The aim of this study is to exploratively assess the efficacy and safety of hydrophilic polyurethane foam in

pressure ulcer patients.

For this purpose, the percentage of completely healed patients and the time to complete healing will be

assessed after applying a study device, Medifoam<sup>®</sup> or Betafoam<sup>®</sup>, for 12 weeks to pressure ulcer patients. In

addition, the pressure ulcer size reduction rate over 12 weeks will be evaluated.

3. Study Design

This is a single-center, randomized, 2-arms, open-label pilot study.

Subjects who consent to the study will be assessed for eligibility with screening tests. Subjects can have a 2-

week screening period.

After screening, subjects who meet the inclusion/exclusion criteria will apply Medifoam® or Betafoam® for

12 weeks, after randomization. Targeted subjects are outpatient clinic or hospitalized patients. Subjects will

make once weekly site visits.

During the treatment period, dressing is performed twice weekly, but additional dressing changes are allowed,

depending on the condition of the pressure ulcer, such as excessive exudates at the study ulcer. Nevertheless,

the frequency of additional dressing is limited to twice daily. On the weekly site visit days, the investigator(or

clinical research coordinator) will change the dressing; on other occasions, the subject or guardian will perform

self-dressing. Subjects who achieve complete healing of the target pressure ulcer within 12 weeks will have

early completion.

Efficacy assessment is conducted for a total of 12 times at a 1-week interval, after the investigational device application (8d, 15d, 22d, 29d, 36d, 43d, 50d, 57d, 64d, 71d, 78d, 85d). At each efficacy assessment, the investigator (or clinical research coordinator) should take a digital photograph of the target pressure ulcer and retain it as a source document.



#### 4. Inclusion/Exclusion Criteria

#### **Inclusion**

- 1) Adults aged at least 19 years old as of the consent date
- 2) Pressure ulcer of the NPUAP(National Pressure Ulcer Advisory Panel) Stage III at screening
- 3) Pressure ulcer size of 3-100 cm<sup>2</sup> at screening
- 4) Written consent provided by the subject or representative (In case a subject has more than one pressure ulcers that meet all inclusion criteria, the largest one is selected as a target lesion.)

#### **Exclusion**

- 1) Any study ulcer of the NPUAP Stage I, II or IV
- 2) Diabetic ulcer or Venous ulcer (or stasis ulcer)
- 3) Past history of surgical treatment within 1 year or irradiation at the target pressure ulcer within 1 year
- 4) Hypersensitivity reaction to this product or povidone-iodine
- 5) Hyperthyroidism or thyroid disorder requiring drug treatment
- 6) Signs of a current underlying systemic infection (sepsis/bacterial infection/tuberculosis) or cellulitis or osteomyelitis
- 7) Type 1 diabetes

8) Current malnutrition

9) Heavy smoker: Current smoking level of ≥1 pack (20 cigarettes)/day of tobacco

10) Drug or alcohol addiction

11) Requirement of immunosuppressants during the study or current chemotherapy or radiotherapy

12) Application of other investigational product/medical device within 1 month prior to the

investigational device application (1d)

13) Pregnant or breastfeeding women

14) Other renal, hepatic, neurological, immunological disorder that may interfere with the wound

healing process, at the discretion of the investigator

5. Discontinuation/Withdrawal and early completion criteria

Discontinuation and withdrawal criteria

In case of meeting the following criteria for study device discontinuation, application of the study device and

the study should be discontinued, and the reason for discontinuation and findings should be recorded in the

Case Report Form.

- Criteria for discontinuation of the study device application

1) Acute reactions (allergy, hypersensitivity reactions, etc.) to the study device

2) It is determined that continuation of the study is difficult due to an accidental intercurrent condition.

3) It is determined that continuation of the study is impossible due to worsening of the pressure ulcer

(Stage 4 or higher).

4) Debridement was performed during the study, after the study device application.

5) Pregnant during the study period

6) It is otherwise determined by the investigator that continued application of the study device is not

appropriate due to reasons such as serious malnutrition, etc.

7) It is determined by the investigator that study participation is not appropriate due to a "serious

adverse event".

"Serious adverse event" is an event, irrespective of a causal relationship with the study device, that is as

follows:

1 Results in death or is life-threatening

② Requires inpatient hospitalization or prolongation of existing hospitalization

SAA-SAP-APX-01 Statistical Analysis Plan Effective Date: 01 AUG 2015

7 of 40

3 Results in persistent or significant disability or dysfunction

4 Results in congenital anomaly or birth defect

(5) Other medically important event as identified by the Investigator

In case of discontinuation due to worsening of a pressure ulcer, the treating physician will ensure safety of the patient with appropriate tests and treatment, equivalent to the case of an adverse event.

#### Early completion criteria

Subjects who achieve complete healing\* of the target pressure ulcer will complete the study early. Subjects who can complete the study early will undergo all tests scheduled for the End-of-Study (85d) visit and then complete the study.

(\* Complete healing: Defined as the condition with the epithelial tissue covering 100% of the study ulcer, no abrasion or ulceration, intact dermis and epidermis.)

#### 6. Statistical Analysis Population

Data obtained from subjects in this study will be analyzed as the SS(Safety Set) and the FAS(Full Analysis set).

1) In the SS(Safety set), data obtained from subjects who were enrolled in the study, had at least 1 application of the study device, and had at least 1 safety assessment will be analyzed.

2) In the FAS(Full analysis set), data obtained from subjects who were enrolled in the study, had at least 1 application of the study device and then had at least 1 available endpoint of main interest review will be included in analysis.

#### 7. Analysis of endpoints

#### 7.1 Efficacy Endpoints

#### (1) Endpoints of main interest

1 Number of patients with complete healing# of ulcer within 12 weeks

: Subjects who achieved complete healing and had early completion or completion at the end of 12

weeks will be included.

- 2) Time to complete healing# of ulcer within 12 weeks
  - : Time to complete healing is calculated as the number of days from baseline (1d).

(# The definition of complete healing: Epithelial tissue covering 100% of the study ulcer, no abrasion or ulceration, intact dermis and epidermis)

- (3) Pressure ulcer size by each time point
- 4 Pressure ulcer size reduction rate based on a scale at each time point

Reduction Rate=

Pressure ulcer size on 1d\* - Pressure ulcer size at each time point from 8d to End-of-Study\*\*

Pressure ulcer size on 1d X 100%

- \* Using a scale-based pressure ulcer area (cm<sup>2</sup>) measured prior to the study device application
- \*\* Using a scale-based pressure ulcer area (cm²) without re-epithelization\*\*\* measured at each time point after the study device application
- (\*\*\*Re-epithelization: New epithelial tissue covering the pressure ulcer, with no exudate, transudate, or avascular tissue)

#### (2) Other endpoints

1 PUSH reduction rate at each time point

- 2 Dressing change frequency during the entire study period
- : Calculated as the additional dressing frequency beyond twice daily
- 3 Number of subjects with early completion due to complete healing during the study
- (4) Incidence of new infections at the pressure ulcer until Week 12 based on the CSSC

Number of subjects with at least 1 new infection\*\* until Week 12,

Infection incidence = after the study device application X 100%

Total number of subjects

(\*\* Infection: Presence of 'Purulent exudates' or 2 or more symptoms of the CSSC. However, for subjects with an infection at baseline, it is defined as development of an additional symptom other than those confirmed at baseline or recurrence of baseline-identified symptoms after being completely healed.)

#### 7.2 Safety Endpoints

The followings will be evaluated for safety assessment.

#### 1) Adverse event

At every visit, review both local adverse events at the target pressure ulcer and other adverse events.

(Local adverse events at the target pressure ulcer: Erythema, edema, itching, flare, rash, others)

#### 2) Vital signs

Vital signs are analyzed by measuring at every visit until study completion. Measured vital signs are blood pressure(), pulse, and body temperature. In addition, body weight is measured at screening, Week 4 and at the End-of-Study visit. Visits conducted outside of the site will not include body weight measurement.

#### 3) Laboratory tests and physical examination

Laboratory tests are conducted at screening and study completion. For physical examination, normal/abnormal status of findings at screening is confirmed, and it is assessed whether the subject is eligible for study participation. Physical examination is also performed at every subsequent visit. Visits conducted outside of the site will not include physical examination.

#### 8. Statistical Methodology by Endpoints

#### **Analysis of Efficacy Endpoints**

#### (1) Analysis of endpoints of main interest

- (1) For subjects achieving complete healing within 12 weeks, present frequency and percentage. Fisher's exact test will be performed to compare Medifoam and Betafoam treatment groups.
- 2 For the time to 100% complete healing, analyze using the Kaplan-Meier method. Time table for subjects to 100% complete healing will be presented and the survival Plot will be shown as a figure. Subjects not achieving 100% complete healing within 12 weeks will not be considered for evaluation for end point of main interest though ulcer size reduction will be evaluated for those subjects.

For the pressure ulcer size by each time point, present the mean, median, min, max and standard

deviation. t-test will be conducted to compare Medifoam and Betafoam, and paired t-test will be

used to see the difference between each post visit and baseline(1d).

4 For the pressure ulcer size reduction rate, present the mean, median, min, max and standard

deviation. t-test will be conducted to compare Medifoam and Betafoam.

(5) For the analysis for efficacy, conduct sub-analyses by use of topicalantibiotics and glucocorticoids

for the pressure ulcer during the study. t-test will be performed to compare Medifoam and Betafoam,

and paired t-test will be used to see the difference between post visits and baseline(1d).

(2) Analysis of other endpoints

For other endpoints, present the mean, median, min, max and standard deviation for the continuous variable

PUSH reduction rate at each time point, and frequency and percentage for categorical variables of Dressing

change frequency, Number of subjects with early completion due to complete healing, and Incidence of new

infections at the pressure ulcer after investigational device application. t-test and paired t-test will be

conducted for PUSH reduction rate while Fisher's exact test will be used to see the difference between

Meidfoam and Betafoam for Dressing change frequency, Number of subjects with early completion , and

Incidence of new infections.

**Analysis of safety endpoints** 

(1) Adverse events

List all adverse events that occurred by group. Record the frequency of adverse events related or unrelated

with the investigational device by group. For the number of adverse events and the percentage of subjects who

had at least 1 adverse event, present the 95% confidence interval in each treatment group. Analyze adverse

events separately for local adverse events at the target pressure ulcer and other adverse events.

(2) Laboratory test findings

For continuous data, present descriptive statistics (mean, standard deviation, median, minimum, maximum) by

group and time point. In addition, tabulate the proportion of normal/abnormal results by time point in each

group.

(3) Vital signs

For continuous variables, present descriptive statistics (mean, standard deviation, median, minimum,

11 of 40

maximum) for the baseline and end-of-study test findings by group and visit time point.

SAA-SAP-APX-01 Statistical Analysis Plan

#### 9. Handling Missing Values

For subjects with a missing value during the study or who are withdrawn from the study prior to study completion, efficacy analysis will be conducted by applying the LOCF(Last observation Carried Forward), only in case such subjects have available endpoints of main interest assessment results after the investigational device application. However, in case of missing values for other endpoints and safety endpoints, raw data will be used for analysis, without applying LOCF.

#### 10. Midterm Analysis

The midterm analysis will not be conducted for this study.

#### 11. Others

#### **Further Consideration**

- In principle, the analysis shall follow the methods presented in Protocol No. BTF16-AP-401 and the general items regarding statistical analysis procedure shall be described.
- For continuous variables, Shapiro-Wilk test with p-value 0.05 will be used for normality test. t-distribution approximation method will be used for Wilcoxon rank sum test.
- Chi-square test will used on half of Fisher's exact test in case when SAS 9.3 cannot handle the amount of test calculation.

## 12. Dummy Table List

| Analysis<br>Criteria/<br>Analysis Set | Table No. | Analysis Variables | Group<br>Variables | Note |
|---|---|---|---|---|
| | 0101 | Disposition of Subjects | ALL | |
| Disposition of<br>Subjects | 0102 | Detailed reports on discontinued subjects | ALL | |
| · | 0103 | Analysis Set | ALL | |
| | 0201 | Gender | V1(Screening) | Medifoam vs.<br>Betafoam |
| | 0201 | Age(Years) | V1(Screening) | Medifoam vs.<br>Betafoam |
| | 0201 | Age(20-29, 30-39, 40-49, 50-59, 60-69, 70 or more) | V1(Screening) | Medifoam vs.<br>Betafoam |
| | 0201 | Body Weight | V1(Screening) | Medifoam vs.<br>Betafoam |
| | 0201 | Height | V1(Screening) | Medifoam vs.<br>Betafoam |
| Demographics | 0201 | Breast Feeding(Female Only) | V1(Screening) | Medifoam vs.<br>Betafoam |
| FAS | 0201 | Possibility of Pregnancy(Female Only) | V1(Screening) | Medifoam vs.<br>Betafoam |
| | 0201 | Reason for not being able to pregnant | V1(Screening) | |
| | 0201 | Countermeasure for pregnancy | V1(Screening) | |
| | 0201 | Alcohol consumption | V1(Screening) | Medifoam vs.<br>Betafoam |
| | 0201 | Nicotine consumption V1(Screeni | | Medifoam vs.<br>Betafoam |
| | 0201 | Urine HCG test results | V1(Screening) | Medifoam vs.<br>Betafoam |
| | 0301 | Pressure Ulcer V1(Screening) | | Medifoam vs.<br>Betafoam |
| | 0302 | Hypersensitivity | V1(Screening) | Medifoam vs.<br>Betafoam |
| | 0303 | Other Medical History(Past/Current) | V1(Screening) | Medifoam vs.<br>Betafoam |
| Medical History<br>FAS | 0304 | Past Medical History (SOC/PT) | V1(Screening) | Medifoam vs.<br>Betafoam |
| | 0305 | Current Medical History (SOC/PT) | V1(Screening) | Medifoam vs. Betafoam |
| | 0306 | Surgical Procedure | V1(Screening) | Medifoam vs. Betafoam |
| | 0307 | List of Surgical Procedure and Indications for subjects who had surgical procedure | V1(Screening) | Medifoam vs. Betafoam |
| Medication | 0401 | Prior/Concomitant Medication(Y/N) | ALL | Medifoam vs. Betafoam |
| History<br>FAS | 0402 | Prior Medication in detail ((Level 1 / Level 3) of WHO ATC) | ALL | Medifoam vs. Betafoam |

| Analysis<br>Criteria/<br>Analysis Set | Table No. | Analysis Variables | Group<br>Variables | Note |
|---|---|---|---|---|
| | 0403 | Concomitant Medication in detail ((Level 1 / Level 3) of WHO ATC) | ALL | Medifoam vs.<br>Betafoam |
| Pressure ulcer assessment at | 0501 | List of Body Parts where Pressure Ulcer occurred | V1(Screening) | Medifoam vs.<br>Betafoam |
| Screening(Visit1) FAS | 0502 | Pressure ulcer size at Screening | V1(Screening) | Medifoam vs.<br>Betafoam |
| | 0601 | Number of patients with complete healing of ulcer within 12 weeks | ALL | Medifoam vs.<br>Betafoam |
| | 0602 | Time taken for subjects to reach complete healing of ulcer within 12 weeks | ALL | Medifoam vs.<br>Betafoam |
| Anahuia af | Figure 0601 | Time to complete healing of ulcer within 12 weeks | ALL | Medifoam vs.<br>Betafoam,<br>Kaplan-Meire Plot |
| Analysis of endpoints of | 0603 | Pressure ulcer size by each time point and change from 1d (Baseline) | ALL | Medifoam vs.<br>Betafoam |
| main interest<br>FAS | 0604 | Pressure ulcer size reduction rate based on scale at each time point | ALL | Medifoam vs.<br>Betafoam |
| | 0605 | Sub-analysis on Pressure ulcer size reduction rate based on scale at each time point by use of topical antibiotics | ALL | Medifoam vs.<br>Betafoam, |
| | 0606 | Sub-analysis on Pressure ulcer size reduction rate based on scale at each time point by use of glucocorticoids | ALL | Medifoam vs.<br>Betafoam |
| | 0701 | PUSH reduction rate at each time point | ALL | Medifoam vs.<br>Betafoam |
| | 0702 | Dressing change frequency during the entire study period for subjects on Medifoam | ALL | Medifoam vs.<br>Betafoam |
| | 0703 | Dressing change frequency during the entire study period for subjects on Betafoam | ALL | Medifoam vs.<br>Betafoam |
| Analysis of | 0704 | Number of subjects with early completion due to complete healing during the study | ALL | Medifoam vs.<br>Betafoam |
| other endpoints<br>FAS | 0705 | Number of subjects by CSSC signs and symptoms per each visit for subjects on Medifoam | ALL | Medifoam vs.<br>Betafoam |
| | 0706 | Number of subjects by CSSC signs and symptoms at each visit for subjects on Betafoam | ALL | Medifoam vs.<br>Betafoam |
| | 0707 | Incidence of new infections at the pressure ulcer until Week 12 based on the CSSC | ALL | |
| Physical<br>Examination<br>Safety | 0801~0813 | Normal(or Abnormal(NCS)/Abnormal(CS)) cross table for Physical Examination | ALL | Medifoam vs.<br>Betafoam<br>McNemar Test |
| Vital Sign | 0901 | Vital Sign Results and Change from Baseline(Temperature) | ALL | Medifoam vs.<br>Betafoam |
| Safety | 0902 | Vital Sign Results and Change from Baseline(SBP, DBP, Pulse) | ALL | Medifoam vs.<br>Betafoam |
| | 1001 | Laboratory Test results and Change from Baseline (Hematology) | ALL | Medifoam vs.<br>Betafoam |
| Laboratory Test<br>Safety | 1002 | Normal(or Abnormal(NCS)/Abnormal(CS)) cross table for Laboratory Test (Hematology) | ALL | Medifoam vs.<br>Betafoam<br>McNemar Test |
| | 1003 | Laboratory Test results and Change from Baseline (Blood Chemistry) | ALL | Medifoam vs.<br>Betafoam |

| Analysis<br>Criteria/<br>Analysis Set | Table No. | Analysis Variables | Group<br>Variables | Note |
|---|---|---|---|---|
| | 1004 | Normal(or Abnormal(NCS)/Abnormal(CS)) cross table for Laboratory Test (Blood Chemistry) | ALL | Medifoam vs.<br>Betafoam<br>McNemar Test |
| | 1101 AE Summary(AE, ADE, SAE, SADE) ALL | | ALL | Medifoam vs.<br>Betafoam |
| | 1102~1105 | Number and Percentage of subjects with (AE, ADE, SAE, SADE ) | ALL | Medifoam vs.<br>Betafoam |
| Adverse Events<br>Safety | 1106~1111 | Incidence rate, Number and frequency of (Local AE, ADE, SAE, SADE) by Severity, SAE, Outcome, Relationship with the clinical device, Action taken with the Device, Seriousness | ALL | Medifoam vs.<br>Betafoam |
| | 1112~1117 | Incidence rate, Number and frequency of (Other AE, ADE, SAE, SADE) by Severity, SAE, Outcome, Relationship with the clinical device, Action taken with the Device, Seriousness | ALL | Medifoam vs.<br>Betafoam |

#### **13. TLFs**

## 1) Disposition of Subjects

## Table 0101 Disposition of Subjects who participated in the study

| | Medifoam | Betafoam | Total |
|---|---|---|---|
| Subjects who signed the Informed Consent form | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) |
| Screening | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) |
| Screening Failure | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) |
| Reason for Screening Failure1 | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) |
| Reason for Screening Failure2 | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) |
| Reason for Screening Failure3 | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) |
| Randomized | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) |
| Reason for Discontinuation 1 | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) |
| Reason for Discontinuation 2 | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) |
| Reason for Discontinuation 3 | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) |
| Subjects who completed the trial (including Early completion) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) |

## Table 0102 Detailed reports on discontinued subjects

| Treatment<br>Group | Screening<br>No. | Randomization<br>No. | Informed<br>Consent<br>Date | Discontinuation<br>Date | Reason for<br>Discontinuation |
|---|---|---|---|---|---|

## Table 0103 Analysis Set

| | Medifoam | Betafoam | Total |
|-----------------------------|------------|------------|------------|
| Randomized | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) |
| Reason1 for Safety excluded | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) |
| Reason2 for Safety excluded | | | |
| Safety Set | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) |
| Reason1 for FAS excluded | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) |
| Reason2 for FAS excluded | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) |
| FAS | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) |

## 2) Demographics Analysis Set: FAS

Table 0201 Demographics

| | T | | T | | |
|---|---|---|---|---|---|
| | | Medifoam | Betafoam | Total | p-value |
| | Male | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | 0.xxxx‡ |
| Gender | Female | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | |
| | Total | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | |
| | N | xx | xx | xx | 0.xxxx* |
| Age | Mean±Std | xx.xx±x.xx | xx.xx±x.xx | xx.xx±x.xx | |
| (Years) | Median | XX.XX | XX.XX | xx.xx | |
| | Min~Max | xx.xx~xx.xx | xx.xx~xx.xx | xx.xx~xx.xx | |
| | 19~29 | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | 0.xxxx‡ |
| | 30~39 | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | |
| A | 40~49 | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | |
| Age<br>(Categorical) | 50~59 | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | |
| (Categorical) | 60~69 | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | |
| | 70< | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | |
| | Total | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | |
| | N | xx | xx | xx | 0.xxxx* |
| Body Weight | Mean±Std | xx.xx±x.xx | xx.xx±x.xx | xx.xx±x.xx | |
| (kg) | Median | XX.XX | XX.XX | xx.xx | |
| | Min~Max | xx.xx~xx.xx | xx.xx~xx.xx | xx.xx~xx.xx | |
| | N | xx | xx | xx | 0.xxxx* |
| Height | Mean±Std | xx.xx±x.xx | xx.xx±x.xx | xx.xx±x.xx | |
| (cm) | Median | xx.xx | xx.xx | xx.xx | |
| | Min~Max | xx.xx~xx.xx | xx.xx~xx.xx | xx.xx~xx.xx | |
| Proact Fooding | Yes | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | 0.xxxx‡ |
| Breast Feeding (Female Only) | No | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | |
| (remale omy) | Total | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | |
| Possibility of | Yes | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | 0.xxxx‡ |
| Pregnancy | No | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | |
| (Yes/No) | Total | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | |
| Reason for not | Menopause 1 year ago | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | |
| being able to get | Hysterectomy/bilateral ovariectomy surgery | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | |
| pregnant | Total | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | |
| | Yes (Condom) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | |
| Countermeasure | Yes (Oral | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | |
| for pregnancy | contraception) | | | AA(AA.XX/0) | |
| .o. pregnancy | Yes (Injectable | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | |
| | contraceptive) | | | 70.(70.00070) | |

| | Yes (Insertable | xx(xx.xx%) | xx(xx.xx%) | , , , , , , | |
|---|---|---|---|---|---|
| | contraceptive) | , , | , | xx(xx.xx%) | |
| | Yes (Intrauterine | xx(xx.xx%) | xx(xx.xx%) | | |
| | contraceptive device) | | | xx(xx.xx%) | |
| | Total | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | |
| Alcohol | Yes | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | 0.xxxx‡ |
| consumption | No | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | |
| Consumption | Total | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | |
| Alcohol | N | xx | xx | xx | 0.xxxx* |
| consumption | Mean±Std | xx.xx±x.xx | xx.xx±x.xx | xx.xx±x.xx | |
| (If yes, alcohol | Median | xx.xx | xx.xx | xx.xx | |
| per week) | Min~Max | xx.xx~xx.xx | xx.xx~xx.xx | xx.xx~xx.xx | |
| Nicotion | Yes | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | 0.xxxx‡ |
| Nicotine | No | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | |
| consumption | Total | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | |
| Nicotine | N | xx | xx | XX | 0.xxxx* |
| consumption(If | Mean±Std | xx.xx±x.xx | xx.xx±x.xx | xx.xx±x.xx | |
| yes, cigarettes | Median | xx.xx | xx.xx | xx.xx | |
| per day) | Min~Max | xx.xx~xx.xx | xx.xx~xx.xx | xx.xx~xx.xx | |
| | Done | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | 0.xxxx‡ |
| Urine HCG Test | Not Done | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | |
| Offile acd lest | Not Applicable | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | |
| | Total | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | |
| Urine Test | Negative | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | 0.xxxx‡ |
| Results | Positive | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | |
| nesuits | Total | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | |

Note) Percentage is based on FAS Set subjects within each column.

Note) \*: t-test, ¥: Wilcoxon rank sum test, ‡: Fisher's exact test

## 3) Medical History

Analysis Set: FAS

Table 0301 Pressure Ulcer

| | | Medifoam | Betafoam | Total | P-value |
|---|---|---|---|---|---|
| | | n(%) | n(%) | n(%) | P-value |
| Prior surgical | Yes | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | 0.xxxx‡ |
| history of target | No | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | |
| ulcer within 1 | Total | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | |
| year | | | | | |
| Prior irradiation | Yes | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | 0.xxxx‡ |
| history of the | No | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | |
| target ulcer | Total | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | |
| within 1 year | | | | | |
| Malnutrition | Yes | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | 0.xxxx‡ |
| Status | No | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | |
| Status | Total | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | |
| | Ambulatory | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | 0.xxxx‡ |
| | Stays sitting only | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | |
| Mobility and | Stays lying only | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | |
| condition | Stays lying and | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | |
| | sitting only | | | | |
| | Total | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | |
| Duration since | N | XX | XX | xx | 0.xxxx* |
| occurrence of | Mean±Std | xx.xx±x.xx | xx.xx±x.xx | xx.xx±x.xx | |
| pressure | Median | xx.xx | xx.xx | xx.xx | |
| ulcer(weeks) | Min~Max | xx.xx~xx.xx | xx.xx~xx.xx | xx.xx~xx.xx | |

<sup>‡:</sup> Fisher's exact test \*: t-test, ¥: Wilcoxon rank sum test

## Table 0302 Hypersensitivity

| | | Medifoam | Betafoam | Total | P-value |
|---------------------|-------|------------|------------|------------|---------|
| | | n(%) | n(%) | n(%) | P-value |
| Hypersensitive to | Yes | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | 0.xxxx‡ |
| povidone-iodine or | No | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | |
| similar medical | Total | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | |
| devices in the past | | | | | |

<sup>‡:</sup> Fisher's exact test

Table 0303 Other medical history and concomitant illness

| | | Medifoam | Betafoam | Total | Divolue |
|---|---|---|---|---|---|
| _ | | n(%) | n(%) | n(%) | P-value |
| Past Medical History | Yes | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | 0.xxxx‡ |
| | No | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | |
| | Total | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | |
| Current Medical | Yes | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | 0.xxxx‡ |
| History | No | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | |
| | Total | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | |

<sup>‡:</sup> Fisher's exact test

#### Table 0304 Past Medical history (SOC/PT\*)

| | | Medifoam | | | | Betafoam | | | Total | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | (N=xx) | | | | (N=xx) | | | (N=xx) | |
| | | n | (%) | freq | n | (%) | freq | N | (%) | freq |
| Total | | XX | (xx.xx) | xx | XX | (xx.xx) | xx | Xx | (xx.xx) | xx |
| SOC | PT | XX | (xx.xx) | XX | XX | (xx.xx) | xx | Xx | (xx.xx) | xx |
| 300 | PT | XX | (xx.xx) | XX | XX | (xx.xx) | XX | Xx | (xx.xx) | xx |

Note ) SOC: System Organ Class, PT: Preferred Term, \* Coded in MedDRA Ver 18.1 or latest version

#### Table 0305 Current Medical history (SOC/PT\*)

| | Medifoam | | | Betafoam | | | Total | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | (N=xx) | | (N=xx) | | | (N=xx) | | |
| | | n | (%) | freq | n | (%) | freq | N | (%) | freq |
| Total | | XX | (xx.xx) | xx | xx | (xx.xx) | xx | Xx | (xx.xx) | xx |
| SOC | PT | XX | (xx.xx) | XX | XX | (xx.xx) | xx | Xx | (xx.xx) | xx |
| 300 | PT | XX | (xx.xx) | XX | XX | (xx.xx) | XX | Xx | (xx.xx) | XX |

Note ) SOC: System Organ Class, PT: Preferred Term, \* Coded in MedDRA Ver 18.1 or latest version

## Table 0306 Surgical Procedure (Yes/No)

| | | Medifoam | Betafoam | Total | P-value |
|--------------------|-------|------------|------------|------------|---------|
| | | n(%) | n(%) | n(%) | P-value |
| | Yes | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | 0.xxxx‡ |
| Surgical Procedure | No | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | |
| _ | Total | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | |

<sup>‡:</sup> Fisher's exact test

Table 0307 List of Surgical Procedure and Indications for subjects who had surgical procedure (Indication/Surgical Procedure)

| | | Medifoam | | | | Betafoam | | | Total | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | (N=xx) | | | (N=xx) | | | (N=xx) | | |
| | | n | (%) | freq | n | (%) | freq | n | (%) | freq |
| Total | | XX | (xx.xx) | XX | XX | (xx.xx) | XX | XX | (xx.xx) | XX |
| Indication | Surgical<br>Procedure | XX | (xx.xx) | XX | xx | (xx.xx) | xx | xx | (xx.xx) | хх |
| maleation | Surgical<br>Procedure | XX | (xx.xx) | XX | XX | (xx.xx) | XX | XX | (xx.xx) | ХХ |

## 4) Medication History

Analysis Set: FAS

Table 0401 Prior/Concomitant Medication

| | | Medifoam | Betafoam | Total | Divolue |
|---|---|---|---|---|---|
| | | n(%) | n(%) | n(%) | P-value |
| | Yes | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | 0.xxxx‡ |
| Prior Medication | No | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | |
| | Total | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | |
| Concomitant | Yes | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | 0.xxxx‡ |
| Concomitant<br>Medication | No | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | |
| iviedication | Total | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | |

<sup>‡:</sup> Fisher's exact test

Table 0402 Prior Medication in detail((Level1/Level3) of WHO ATC\*)

| | | Med | difoam | Bet | afoam | To | otal |
|--------|--------|-----|---------|-----|---------|----|---------|
| | | n | (%) | n | (%) | n | (%) |
| Total | | XX | (xx.xx) | XX | (xx.xx) | XX | (xx.xx) |
| Level1 | Level3 | XX | (xx.xx) | XX | (xx.xx) | XX | (xx.xx) |
| LCVEIT | Level3 | XX | (xx.xx) | XX | (xx.xx) | XX | (xx.xx) |

Note) \* Coded in WHO ATC Class

## Table 0403 Concomitant Medication in detail ((Level 1/ Level 3) of WHO ATC\*)

| | | Medifoam | | | Betafoam | | | Total | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | n | (%) | freq | n | (%) | freq | N | (%) | freq |
| Total | | XX | (xx.xx) | xx | XX | (xx.xx) | xx | XX | (xx.xx) | xx |
| Level1 | Level3 | XX | (xx.xx) | xx | XX | (xx.xx) | XX | XX | (xx.xx) | xx |
| Levell | Level3 | XX | (xx.xx) | XX | XX | (xx.xx) | XX | XX | (xx.xx) | XX |

Note) Percentage is based on FAS Set subjects within each column.

Note) \* Coded in WHO ATC Class

## 5) Pressure ulcer assessment at Screening(Visit1)

Table 0501 List of body parts where pressure ulcer occurred

| | Medifoam | Betafoam | Total |
|-----------|----------|----------|-------|
| Body Part | n | n | n |
| Location1 | XX | XX | XX |
| Location2 | XX | xx | xx |
| Location3 | XX | xx | xx |
| Location4 | XX | xx | xx |
| | XX | XX | xx |
| Total | XX | xx | xx |

Table 0502 Pressure ulcer size at Screening

| Measureme | nt | Medifoam | Betafoam | Total | P-value |
|-------------|----------|-------------|-------------|-------------|---------|
| | N | xx | xx | xx | 0.xxxx* |
| Length(cm) | Mean±Std | xx.xx±x.xx | xx.xx±x.xx | xx.xx±x.xx | |
| | Median | XX.XX | XX.XX | xx.xx | |
| | Min~Max | xx.xx~xx.xx | xx.xx~xx.xx | xx.xx~xx.xx | |
| | N | xx | xx | XX | 0.xxxx* |
| \\/;d+b/am\ | Mean±Std | xx.xx±x.xx | xx.xx±x.xx | xx.xx±x.xx | |
| Width(cm) | Median | XX.XX | XX.XX | xx.xx | |
| | Min~Max | xx.xx~xx.xx | xx.xx~xx.xx | xx.xx~xx.xx | |

## 6) Analysis of endpoints of main interest

Analysis Set: FAS

Table 0601 Number of patients with complete healing of ulcer within 12 weeks

| | | | Betafoam | Total | P-value |
|--------------------|-------|------------|------------|------------|---------|
| | | | n(%) | n(%) | r-value |
| Complete healing | Yes | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | 0.xxxx‡ |
| of ulcer within 12 | No | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | |
| weeks | Total | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | |

<sup>‡:</sup> Fisher's exact test

## Table 0602Time taken for subjects to reach complete healing of ulcer within 12 weeks(in days)

| | | Medifoam | Betafoam | Total | P-value |
|--------------|----------|-------------|-------------|-------------|---------|
| | N | xx | xx | xx | 0.xxxx* |
| Time(days) | Mean±Std | xx.xx±x.xx | xx.xx±x.xx | xx.xx±x.xx | |
| ·····c(dd/5) | Median | xx.xx | xx.xx | xx.xx | |
| | Min~Max | xx.xx~xx.xx | xx.xx~xx.xx | xx.xx~xx.xx | |

Note) \*: t-test, \(\forall : \text{Wilcoxon rank sum test}\)

Figure 0601 Time to complete healing of ulcer within 12 weeks



Table 0603 Pressure ulcer size by each time point and change from 1d (baseline)

| Time points | | Medifoam | Betafoam | Total | P-value |
|---|---|---|---|---|---|
| | N | xx | XX | XX | 0.xxxx* |
| \/ici+2/1d\ | Mean±Std | xx.xx±x.xx | xx.xx±x.xx | xx.xx±x.xx | |
| Visit2(1d) | Median | xx.xx | XX.XX | xx.xx | |
| | Min~Max | xx.xx~xx.xx | xx.xx~xx.xx | xx.xx~xx.xx | |
| | N | XX | XX | XX | 0.xxxx* |
| \/ici+2/0d±1d\ | Mean±Std | xx.xx±x.xx | xx.xx±x.xx | xx.xx±x.xx | |
| Visit3(8d±1d) | Median | xx.xx | XX.XX | xx.xx | |
| | Min~Max | xx.xx~xx.xx | xx.xx~xx.xx | xx.xx~xx.xx | |
| Visit4~Visit14 | | (M | iddle Part omitte | ed) | |

Note) \*: t-test, \(\forall : \text{Wilcoxon rank sum test}\)

Table 0604 Pressure ulcer size reduction rate based on scale at each time point

| Time points | | Medifoam | Betafoam | Total | P-value |
|---|---|---|---|---|---|
| | | n(%) | n(%) | n(%) | r-value |
| | N | XX | XX | XX | 0.xxxx* |
| | Mean±Std | xx.xx±x.xx | xx.xx±x.xx | xx.xx±x.xx | |
| Visit3(8d±1d) | Median | xx.xx | XX.XX | XX.XX | |
| | Min~Max | xx.xx~xx.xx | xx.xx~xx.xx | xx.xx~xx.xx | |
| | P-value(within) | 0.xxxx# | | | |

| Visit4~Visit13 | (Middle Part omitted) | | | | |
|---|---|---|---|---|---|
| | N | XX | XX | XX | 0.xxxx* |
| | Mean±Std | xx.xx±x.xx | xx.xx±x.xx | xx.xx±x.xx | |
| Visit14(85d±2d) | Median | XX.XX | XX.XX | XX.XX | |
| | Min~Max | xx.xx~xx.xx | xx.xx~xx.xx | xx.xx~xx.xx | |
| | P-value(within) | 0.xxxx# | | | |

Note) \*: t-test, ¥: Wilcoxon rank sum test #: Paired t-test, \$: Wilcoxon signed rank test

Table 0605 Sub-analysis on Pressure ulcer size reduction rate based on scale at each time point by Use of topical antibiotics

| Use of Topical antibiotics | Time | points | Medifoam | Betafoam | Total | P-value |
|---|---|---|---|---|---|---|
| | | N | xx | XX | XX | 0.xxxx* |
| | \/;c;+2/0d+1d\ | Mean±Std | xx.xx±x.xx | xx.xx±x.xx | xx.xx±x.xx | |
| | Visit3(8d±1d) | Median | xx.xx | xx.xx | XX.XX | |
| Topical | | Min~Max | xx.xx~xx.xx | xx.xx~xx.xx | xx.xx~xx.xx | |
| antibiotics | Visit4~Visit13 | | (Mido | dle Part Omitte | d) | |
| used | | N | xx | XX | xx | 0.xxxx* |
| | \/'-':44/05 d.2d\ | Mean±Std | xx.xx±x.xx | xx.xx±x.xx | xx.xx±x.xx | |
| | Visit14(85d±2d) | Median | xx.xx | xx.xx | xx.xx | |
| | | Min~Max | xx.xx~xx.xx | xx.xx~xx.xx | xx.xx~xx.xx | |
| | | N | xx | xx | XX | 0.xxxx* |
| | \/;c;+2/0d+1d\ | Mean±Std | xx.xx±x.xx | xx.xx±x.xx | xx.xx±x.xx | |
| | Visit3(8d±1d) | Median | xx.xx | xx.xx | xx.xx | |
| Topical | | Min~Max | xx.xx~xx.xx | xx.xx~xx.xx | xx.xx~xx.xx | |
| antibiotics | Visit4~Visit13 | | (Midd | dle Part Omitte | d) | |
| Not used | | N | xx | xx | XX | 0.xxxx* |
| | \/;c;+1.4/0Fd+2d\ | Mean±Std | xx.xx±x.xx | xx.xx±x.xx | xx.xx±x.xx | |
| | Visit14(85d±2d) | Median | xx.xx | xx.xx | xx.xx | |
| | | Min~Max | xx.xx~xx.xx | xx.xx~xx.xx | xx.xx~xx.xx | |

Note) \*: t-test, ¥: Wilcoxon rank sum test

Table 0606 Sub-analysis on Pressure ulcer size reduction rate based on scale at each time point by Use of glucocorticoids

| Use of glucocorticoids | Time po | ints | Medifoam | Betafoam | Total | P-value |
|---|---|---|---|---|---|---|
| | | N | xx | xx | xx | 0.xxxx* |
| | \/;c;+2/0d+1d\ | Mean±Std | xx.xx±x.xx | xx.xx±x.xx | xx.xx±x.xx | |
| | Visit3(8d±1d) | Median | xx.xx | xx.xx | xx.xx | |
| Chronomtinoida | | Min~Max | xx.xx~xx.xx | xx.xx~xx.xx | xx.xx~xx.xx | |
| Glucocorticoids | Visit4~Visit13 | | (Mido | lle Part Omitt | ed) | |
| used | | N | xx | xx | xx | 0.xxxx* |
| | Visit14(85d±2d) | Mean±Std | xx.xx±x.xx | xx.xx±x.xx | xx.xx±x.xx | |
| | | Median | xx.xx | xx.xx | xx.xx | |
| | | Min~Max | xx.xx~xx.xx | xx.xx~xx.xx | xx.xx~xx.xx | |
| | | N | xx | xx | XX | 0.xxxx* |
| | V''-'12/0-l14-lV | Mean±Std | xx.xx±x.xx | xx.xx±x.xx | xx.xx±x.xx | |
| | Visit3(8d±1d) | Median | xx.xx | xx.xx | xx.xx | |
| Chusasartiaaids | | Min~Max | xx.xx~xx.xx | xx.xx~xx.xx | xx.xx~xx.xx | |
| Glucocorticoids | Visit4~Visit13 | | (Mido | lle Part Omitt | ed) | |
| Not used | | N | xx | xx | XX | 0.xxxx* |
| | \/;c;+1.4/0F.d+2.d\ | Mean±Std | xx.xx±x.xx | xx.xx±x.xx | xx.xx±x.xx | |
| | Visit14(85d±2d) | Median | xx.xx | xx.xx | xx.xx | |
| | | Min~Max | xx.xx~xx.xx | xx.xx~xx.xx | xx.xx~xx.xx | |

Note) \*: t-test, ¥: Wilcoxon rank sum test

## 7) Analysis of Other endpoints

Analysis Set: FAS

Table 0701 PUSH reduction rate at each time point compared to baseline

| Time points | | Medifoam | Betafoam | Total | P-value |
|---|---|---|---|---|---|
| | N | XX | XX | XX | 0.xxxx* |
| | Mean±Std | xx.xx±x.xx | xx.xx±x.xx | xx.xx±x.xx | |
| Visit3(8d±1d) | Median | xx.xx | xx.xx | xx.xx | |
| VISItS(8u±1u) | Min~Max | xx.xx~xx.xx | xx.xx~xx.xx | xx.xx~xx.xx | |
| | P- | 0.xxxx | | | |
| | value(within) | | | | |
| Visit4~Visit13 | | (Mid | dle Part Omitt | ed) | |
| | N | XX | XX | XX | 0.xxxx* |
| | Mean±Std | xx.xx±x.xx | xx.xx±x.xx | xx.xx±x.xx | |
| \/ici+14/9Ed+2d\ | Median | xx.xx | xx.xx | xx.xx | |
| Visit14(85d±2d) | Min~Max | xx.xx~xx.xx | xx.xx~xx.xx | xx.xx~xx.xx | |
| | P- | 0.xxxx | | | |
| | value(within) | | | | |

Note) \*: t-test, ¥: Wilcoxon rank sum test

Table 0702 Dressing change frequency per week during the entire study period for subjects on Medifoam

| | | Medifoam | | |
|---|---|---|---|---|
| | | Vis | sits | |
| Number of Dressing Change per week | Visit3 | Visit4 | | Visit14 |
| None | N | N | N | N |
| One time | N | N | N | N |
| Two times | N | N | N | N |
| Three times | N | N | N | N |
| Four or more times | N | N | N | N |
| Total | N | N | N | N |

Table 0703 Dressing change frequency per week during the entire study period for subjects on Betafoam

<sup>\*</sup>Same as 0702

| | | Medifoam | Betafoam | Total | P-value |
|------------------|-------|------------|------------|------------|---------|
| | | n(%) | n(%) | n(%) | 1 Value |
| Early completion | Yes | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | 0.xxxx‡ |
| due to complete | No | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | |
| healing | Total | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | |

Note) ‡: Fisher's exact test

# Table 0705 Number of subjects with CSSC signs and symptoms at each visit for subjects on Medifoam

| | Medifoam | | | |
|--------------------------------------|----------|--------|---|---------|
| CSSC signs and symptoms | Visit2 | Visit3 | | Visit14 |
| Increasing pain in the ulcer area | N | N | N | N |
| Can't detect pain in ulcer area | N | N | N | N |
| Have less pain now than in the past | N | N | N | N |
| Intensity of pain remained the same | N | N | N | N |
| More ulcer pain now than in the past | N | N | N | N |
| Erythema | N | N | N | N |
| Edema | N | N | N | N |
| Heat | N | N | N | N |
| Purulent exudates | N | N | N | N |
| Sanguinous exudates | N | N | N | N |
| Serous exudates | N | N | N | N |
| Delayed healing of the ulcer | N | N | N | N |
| Discoloration of granulation tissue | N | N | N | N |
| Friable granulation tissue | N | N | N | N |
| Pocketing at base of wound | N | N | N | N |
| Foul odor | N | N | N | N |
| Wound breakdown | N | N | N | N |
| Total | N | N | N | N |

Table 0706 Number of subjects with CSSC signs and symptoms at each visit for subjects on Betafoam \*Same as Table 0705

Table 0707 Incidence of new infections at the pressure ulcer until Week 12 based on the CSSC

| Treatment | n | 95% C.I. of | F | Total |
|-----------|------------------|----------------|-----------|-------|
| group | (Incidence rate) | Incidence rate | Frequency | Total |

| Medifoam | x(x.xx%) | (x.xx,x.xx) | XX | XX |
|----------|----------|-------------|----|----|
| Betafoam | x(x.xx%) | (x.xx,x.xx) | XX | XX |

#### 8) Physical Examination

Analysis Set: Safety

Table 0801 Normal or Abnormal (NCS)/Abnormal(CS)) cross table for Physical Examination (Visit 1 vs. Visit 2)

| | | | | | | | Visit | 2(1d) | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| \/:a:±1/Ca | | Medifoam | | | | | | Betafoam | | | | | |
| VISITT(SC | reening) | Normal Al | | Abno | Abnormal | | Total | | Normal | | Abnormal | | tal |
| | | N | (%) | N | (%) | N | (%) | N | (%) | N | (%) | N | (%) |
| Variables | Normal | xx | Xx<br>(xx.xx) | XX | xx<br>(xx.xx) | XX | xx<br>(xx.xx) | xx | xx<br>(xx.xx) | XX | xx<br>(xx.xx) | XX | xx<br>(xx.xx) |
| | Abnormal | xx | Xx<br>(xx.xx) | xx | xx<br>(xx.xx) | хх | xx<br>(xx.xx) | хх | xx<br>(xx.xx) | хх | xx<br>(xx.xx) | xx | xx<br>(xx.xx) |
| | Total | хх | Xx<br>(xx.xx) | xx | xx<br>(xx.xx) | хх | xx<br>(xx.xx) | xx | xx<br>(xx.xx) | хх | xx<br>(xx.xx) | xx | (xx.xx) |
| P-value | | 0.xxxx | | | | | | 0.xxxx | | | | | |
| | Rest Variables are omitted in TLF | | | | | | | | | | | | |

Note) Normal includes normal and NCS, while abnormal refers to CS.

Note) p-value: McNemar test

Table 0702 Normal (or Abnormal (NCS)/Abnormal(CS) cross table for Physical Examination (Visit 1 vs. Visit 3)

\*Same as Table 0801

Table 0803 Normal or Abnormal (NCS)/Abnormal(CS) cross table for Physical Examination (Visit 1 vs. Visit 4)

\*Same as Table 0801

Table 0804 Normal or Abnormal (NCS)/Abnormal(CS) cross table for Physical Examination (Visit 1 vs. Visit 5)

\*Same as Table 0801

Table 0805 Normal or Abnormal (NCS)/Abnormal(CS) cross table for Physical Examination (Visit 1 vs. Visit 6)

\*Same as Table 0801

Table 0806 Normal or Abnormal (NCS)/Abnormal(CS) cross table for Physical Examination (Visit 1 vs. Visit 7)

\*Same as Table 0801

Table 0807 Normal or Abnormal (NCS)/Abnormal(CS) cross table for Physical Examination (Visit 1 vs. Visit 8)

\*Same as Table 0801

Table 0808 Normal or Abnormal (NCS)/Abnormal(CS) cross table for Physical Examination (Visit 1 vs. Visit 9)

\*Same as Table 0801

Table 0809 Normal or Abnormal (NCS)/Abnormal(CS) cross table for Physical Examination (Visit 1 vs. Visit 10)

\*Same as Table 0801

Table 0810 Normal or Abnormal (NCS)/Abnormal(CS) cross table for Physical Examination (Visit 1 vs. Visit 11)

\*Same as Table 0801

Table 0811 Normal or Abnormal (NCS)/Abnormal(CS) cross table for Physical Examination (Visit 1 vs. Visit 12)

\*Same as Table 0801

Table 0812 Normal or Abnormal (NCS)/Abnormal(CS) cross table for Physical Examination (Visit 1 vs. Visit 13)

\*Same as Table 0801

Table 0813 Normal or Abnormal (NCS)/Abnormal(CS) cross table for Physical Examination (Visit 1 vs. Visit 14)

\*Same as Table 0801

## 9) Vital Sign

Analysis Set: Safety

Table 0901 Vital Sign Results and Change from Baseline (Temperature)

| Time points | | Medifoam | Betafoam | Total | P-value |
|---|---|---|---|---|---|
| | N | XX | XX | XX | 0.xxxx* |
| \/isi+1/Corooning\ | Mean±Std | xx.xx±x.xx | xx.xx±x.xx | xx.xx±x.xx | |
| Visit1(Screening) | Median | xx.xx | xx.xx | xx.xx | |
| | Min~Max | xx.xx~xx.xx | xx.xx~xx.xx | xx.xx~xx.xx | |
| | N | XX | XX | XX | 0.xxxx* |
| \/;<;+2/0d+1d\ | Mean±Std | xx.xx±x.xx | xx.xx±x.xx | xx.xx±x.xx | |
| Visit3(8d±1d) | Median | xx.xx | xx.xx | xx.xx | |
| | Min~Max | xx.xx~xx.xx | xx.xx~xx.xx | xx.xx~xx.xx | |
| Visit4~Visit13 | | (M | iddle Part Omitte | ed) | |
| | N | XX | XX | XX | 0.xxxx* |
| \/:a:+1.4/0F.d +2.d\ | Mean±Std | xx.xx±x.xx | xx.xx±x.xx | xx.xx±x.xx | |
| Visit14(85d±2d) | Median | xx.xx | xx.xx | xx.xx | |
| | Min~Max | xx.xx~xx.xx | xx.xx~xx.xx | xx.xx~xx.xx | |
| | N | XX | XX | XX | 0.xxxx* |
| | Mean±Std | xx.xx±x.xx | xx.xx±x.xx | xx.xx±x.xx | |
| \/ici+2 \/ici+1 | Median | xx.xx | xx.xx | xx.xx | |
| Visit3-Visit1 | Min~Max | xx.xx~xx.xx | xx.xx~xx.xx | xx.xx~xx.xx | |
| | p- | 0.xxxx <sup>#</sup> | | | |
| | value(within) | | | | |
| [Visit4-Visit1]~ | | / / / / | iddle Part Omitte | ٠٨١ | |
| [Visit13-Visit1] | | (۱۷۱ | iddle Part Offitte | eu) | |
| | N | XX | XX | XX | 0.xxxx* |
| | Mean±Std | xx.xx±x.xx | xx.xx±x.xx | xx.xx±x.xx | |
| Visit14-Visit1 | Median | xx.xx | XX.XX | xx.xx | |
| VISIL14-VISIL1 | Min~Max | xx.xx~xx.xx | xx.xx~xx.xx | xx.xx~xx.xx | |
| | p- | 0.xxxx <sup>#</sup> | | | |
| | value(within) | | | | |

Note) \*: t-test, ¥: Wilcoxon rank sum test, #: Paired t-test, \$: Wilcoxon signed rank test

Table 0902 Vital Sign Results and Change from Baseline (SBP, DBP, Pulse)

| Variables | Time points | | Medifoam | Betafoam | Total | P-value |
|---|---|---|---|---|---|---|
| | | N | XX | xx | xx | 0.xxxx* |
| | \/:a:+1/Caraaning\ | Mean±Std | xx.xx±x.xx | xx.xx±x.xx | xx.xx±x.xx | |
| | Visit1(Screening) | Median | xx.xx | xx.xx | xx.xx | |
| | | Min~Max | xx.xx~xx.xx | xx.xx~xx.xx | xx.xx~xx.xx | |
| | | N | XX | xx | xx | 0.xxxx* |
| | \/:a:+3/0d+1d\ | Mean±Std | xx.xx±x.xx | xx.xx±x.xx | xx.xx±x.xx | |
| | Visit3(8d±1d) | Median | xx.xx | xx.xx | xx.xx | |
| | | Min~Max | xx.xx~xx.xx | xx.xx~xx.xx | xx.xx~xx.xx | |
| | Visit4~Visit13 | | (Midd | le Part Omitted | ) | |
| | | N | XX | XX | XX | 0.xxxx* |
| | \/;c;+1.4/9Fd+2d\ | Mean±Std | xx.xx±x.xx | xx.xx±x.xx | xx.xx±x.xx | |
| | Visit14(85d±2d) | Median | xx.xx | xx.xx | xx.xx | |
| SBP | | Min~Max | xx.xx~xx.xx | xx.xx~xx.xx | xx.xx~xx.xx | |
| SBP | | N | XX | XX | XX | 0.xxxx* |
| SBP | | Mean±Std | xx.xx±x.xx | xx.xx±x.xx | xx.xx±x.xx | |
| | Visit3-Visit1 | Median | xx.xx | xx.xx | xx.xx | |
| | AISIT2-AISITT | Min~Max | xx.xx~xx.xx | xx.xx~xx.xx | xx.xx~xx.xx | |
| | | р- | 0.xxxx <sup>#</sup> | | | |
| | | value(within) | | | | |
| | [Visit4-Visit1]~ | | (Midd) | le Part Omitted | ١ | |
| | [Visit13-Visit1] | | (IVIIdul | | )··· | |
| | | N | XX | XX | xx | 0.xxxx* |
| | | Mean±Std | xx.xx±x.xx | xx.xx±x.xx | xx.xx±x.xx | |
| | Visit14-Visit1 | Median | xx.xx | xx.xx | xx.xx | |
| | A121fT#-A121fT | Min~Max | xx.xx~xx.xx | xx.xx~xx.xx | xx.xx~xx.xx | |
| | | р- | 0.xxxx <sup>#</sup> | | | |
| | | value(within) | | | | |
| | D | BP and Pulse sed | ctions are omit | ted in TLF | | |

Note) \*: t-test, ¥: Wilcoxon rank sum test, #: Paired t-test, \$: Wilcoxon signed rank test

10) Laboratory Test

Analysis Set: Safety

Table 1001 Laboratory Test results and Change from Baseline (Hematology)

| Variables | Time points | | Medifoam | Betafoam | Total | P-value |
|---|---|---|---|---|---|---|
| | | N | XX | XX | XX | 0.xxxx* |
| | Visit1/Scrooning) | Mean±Std | xx.xx±x.xx | xx.xx±x.xx | xx.xx±x.xx | |
| | Visit1(Screening) | Median | xx.xx | xx.xx | xx.xx | |
| | | Min~Max | xx.xx~xx.xx | xx.xx~xx.xx | xx.xx~xx.xx | |
| | | N | xx | XX | xx | 0.xxxx* |
| WBC | Visit14(85d±2d) | Mean±Std | xx.xx±x.xx | xx.xx±x.xx | xx.xx±x.xx | |
| VVBC | | Median | xx.xx | xx.xx | xx.xx | |
| | | Min~Max | xx.xx~xx.xx | xx.xx~xx.xx | xx.xx~xx.xx | |
| | | N | XX | XX | XX | 0.xxxx* |
| | Visit14-Visit1 | Mean±Std | xx.xx±x.xx | xx.xx±x.xx | xx.xx±x.xx | |
| | VISIL14-VISIL1 | Median | xx.xx | xx.xx | xx.xx | |
| | | Min~Max | xx.xx~xx.xx | xx.xx~xx.xx | xx.xx~xx.xx | |
| | Rest Variables are omitted in TLF | | | | | |

Note) \*: t-test, ¥: Wilcoxon rank sum test, #: Paired t-test, \$: Wilcoxon signed rank test

## Table 1002 Normal or Abnormal (NCS)/Abnormal(CS) cross table for Laboratory Test (Hematology)

| | | | | | | ١ | isit14(85 | d±2d) | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| \/:a:±1/6 | | Medifoam | | | | | Betafoam | | | | | | |
| VISITT(S | Visit1(Screening) | | Normal | | Abnormal | | Total | Normal | | Abnormal | | | Total |
| | | N | (%) | N | (%) | N | (%) | N | (%) | N | (%) | N | (%) |
| WBC | Normal | xx | Xx<br>(xx.xx) | xx | xx<br>(xx.xx) | xx | xx<br>(xx.xx) | xx | xx<br>(xx.xx) | xx | xx<br>(xx.xx) | xx | xx<br>(xx.xx) |
| | Abnormal | xx | Xx<br>(xx.xx) | xx | xx<br>(xx.xx) | хх | xx<br>(xx.xx) | xx | xx<br>(xx.xx) | xx | xx<br>(xx.xx) | xx | xx<br>(xx.xx) |
| | Total | | Xx<br>(xx.xx) | xx | xx<br>(xx.xx) | xx | xx<br>(xx.xx) | xx | xx<br>(xx.xx) | xx | xx<br>(xx.xx) | xx | (xx.xx) |
| P-value | | 0.xxxx | | | | | | 0.xxxx | | | | | |
| | Rest Variables are omitted in TLF | | | | | | | | | | | | |

Note) Normal includes normal and NCS, while abnormal refers to CS.

Note) p-value: McNemar test

Table 1003 Laboratory Test results and Change from Baseline (Blood Chemistry)

| Variables | Time points | | Medifoam | Betafoam | Total | P-value |
|---|---|---|---|---|---|---|
| | | N | XX | XX | XX | 0.xxxx* |
| | Visit1(Screening) | Mean±Std | xx.xx±x.xx | xx.xx±x.xx | xx.xx±x.xx | |
| | visit1(screening) | Median | xx.xx | xx.xx | xx.xx | |
| | | Min~Max | xx.xx~xx.xx | xx.xx~xx.xx | xx.xx~xx.xx | |
| | | N | XX | XX | XX | 0.xxxx* |
| ALP | Visit14(85d±2d) | Mean±Std | xx.xx±x.xx | xx.xx±x.xx | xx.xx±x.xx | |
| ALP | | Median | xx.xx | xx.xx | xx.xx | |
| | | Min~Max | xx.xx~xx.xx | xx.xx~xx.xx | xx.xx~xx.xx | |
| | | N | XX | XX | XX | 0.xxxx* |
| | Visit14-Visit1 | Mean±Std | xx.xx±x.xx | xx.xx±x.xx | xx.xx±x.xx | |
| | VISIL14-VISIL1 | Median | xx.xx | xx.xx | xx.xx | |
| | | Min~Max | xx.xx~xx.xx | xx.xx~xx.xx | xx.xx~xx.xx | |
| | | Rest Variable | s are omitted i | n TLF | | |

Note) \*: t-test, ¥: Wilcoxon rank sum test, #: Paired t-test, \$: Wilcoxon signed rank test

Table 1004 Normal or Abnormal (NCS)/Abnormal(CS) cross table for Laboratory Test (Blood Chemistry)

| | | | | | | | Visit14( | 85d±2d) | ) | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| ١ | Visit1 | Medifoam | | | | | Betafoam | | | | | | |
| (Screening) | | Normal | | Abnormal | | Total | | Normal | | Abnormal | | | Total |
| | | N | (%) | N | (%) | N | (%) | N | (%) | N | (%) | N | (%) |
| ALP | ALP Normal | | Xx<br>(xx.xx) | xx | xx<br>(xx.xx) | xx | xx<br>(xx.xx) | xx | xx<br>(xx.xx) | хх | xx<br>(xx.xx) | xx | xx<br>(xx.xx) |
| | Abnormal | xx | Xx<br>(xx.xx) | xx | xx<br>(xx.xx) | xx | xx<br>(xx.xx) | xx | xx<br>(xx.xx) | хх | xx<br>(xx.xx) | xx | xx<br>(xx.xx) |
| | Total | xx | Xx<br>(xx.xx) | xx | xx<br>(xx.xx) | xx | xx<br>(xx.xx) | xx | xx<br>(xx.xx) | хх | xx<br>(xx.xx) | хх | (xx.xx) |
| P-<br>value | | 0.xxxx | | | | | | 0.xxxx | | | | | |
| | Rest Variables are omitted in TLF | | | | | | | | | | | | |

Note1) Normal includes normal and NCS, while abnormal refers to CS.

Note2) p-value: McNemar test

# 11) Adverse Events Analysis Set: Safety

Table 1101 AE Summary (AE, ADE, SAE, SADE)

| AE Type | Adverse Event | Treatment | n<br>(Incidence<br>rate) | 95% C.I. of<br>Incidence<br>rate | Frequency | Total | P-value |
|---|---|---|---|---|---|---|---|
| | | Medifoam | x(x.xx%) | (x.xx,x.xx) | XX | XX | 0.xxxx‡ |
| | AE | Betafoam | x(x.xx%) | (x.xx,x.xx) | XX | XX | |
| | | Total | x(x.xx%) | (x.xx,x.xx) | xx | XX | |
| | | Medifoam | x(x.xx%) | (x.xx,x.xx) | XX | XX | 0.xxxx‡ |
| | ADE | Betafoam | x(x.xx%) | (x.xx,x.xx) | XX | XX | |
| Local | | Total | x(x.xx%) | (x.xx,x.xx) | XX | XX | |
| Local | | Medifoam | x(x.xx%) | (x.xx,x.xx) | XX | XX | 0.xxxx‡ |
| | SAE | Betafoam | x(x.xx%) | (x.xx,x.xx) | xx | XX | |
| | | Total | x(x.xx%) | (x.xx,x.xx) | XX | XX | |
| | | Medifoam | x(x.xx%) | (x.xx,x.xx) | XX | XX | 0.xxxx‡ |
| | SADE | Betafoam | x(x.xx%) | (x.xx,x.xx) | XX | XX | |
| | | Total | x(x.xx%) | (x.xx,x.xx) | XX | XX | |
| | | Medifoam | x(x.xx%) | (x.xx,x.xx) | XX | XX | 0.xxxx‡ |
| | AE | Betafoam | x(x.xx%) | (x.xx,x.xx) | XX | XX | |
| | | Total | x(x.xx%) | (x.xx,x.xx) | xx | XX | |
| | | Medifoam | x(x.xx%) | (x.xx,x.xx) | XX | XX | 0.xxxx‡ |
| | ADE | Betafoam | x(x.xx%) | (x.xx,x.xx) | XX | XX | |
| Other | | Total | x(x.xx%) | (x.xx,x.xx) | XX | XX | |
| Other | | Medifoam | x(x.xx%) | (x.xx,x.xx) | XX | xx | 0.xxxx‡ |
| | SAE | Betafoam | x(x.xx%) | (x.xx,x.xx) | XX | XX | |
| | | Total | x(x.xx%) | (x.xx,x.xx) | XX | XX | |
| | | Medifoam | x(x.xx%) | (x.xx,x.xx) | xx | XX | 0.xxxx‡ |
| | SADE | Betafoam | x(x.xx%) | (x.xx,x.xx) | xx | XX | |
| | | Total | x(x.xx%) | (x.xx,x.xx) | XX | XX | |

Note) ‡: Fisher's exact test

Table 1102 Number and Percentage of subjects with AE (SOC/PT\*)

| | E Tupo | | | Medifoan | n | | Betafoam | | | Total | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | E Type | | n | (%) | freq | n | (%) | freq | n | (%) | freq |
| | Total | | XX | (xx.xx) | XX | XX | (xx.xx) | XX | XX | (xx.xx) | XX |
| Local | SOC | PT | XX | (xx.xx) | XX | XX | (xx.xx) | XX | XX | (xx.xx) | XX |
| | 300 | PT | XX | (xx.xx) | XX | XX | (xx.xx) | XX | XX | (xx.xx) | XX |
| | Total | | XX | (xx.xx) | XX | XX | (xx.xx) | XX | XX | (xx.xx) | XX |
| Other | SOC | PT | XX | (xx.xx) | XX | XX | (xx.xx) | XX | XX | (xx.xx) | XX |
| | 300 | PT | XX | (xx.xx) | XX | XX | (xx.xx) | XX | XX | (xx.xx) | XX |

Note)\* SOC: System Organ Class, PT: Preferred Term, \* Coded in MedDRA Ver 18.1 or the latest version

Table 1103 Number and Percentage of subjects with ADE (SOC/PT)

Table 1104 Number and Percentage of subjects with SAE (SOC/PT)

Table 1105 Number and Percentage of subjects with SADE (SOC/PT)

Table 1106 Incidence rate, number and frequency of Local AE by Severity

| Treatment | Soverity | n | 95% C.I. of | Fraguancy | Total |
|---|---|---|---|---|---|
| Group | Severity | (Incidence rate) | Incidence rate | Frequency | Total |
| | Mild | x(x.xx%) | (x.xx,x.xx) | xx | XX |
| Medifoam | Moderate | x(x.xx%) | (x.xx,x.xx) | xx | XX |
| iviediloaiii | Severe | x(x.xx%) | (x.xx,x.xx) | xx | xx |
| | Total | x(x.xx%) | (x.xx,x.xx) | xx | XX |
| | Mild | x(x.xx%) | (x.xx,x.xx) | XX | XX |
| Betafoam | Moderate | x(x.xx%) | (x.xx,x.xx) | XX | XX |
| Detaioani | Severe | x(x.xx%) | (x.xx,x.xx) | xx | xx |
| | Total | x(x.xx%) | (x.xx,x.xx) | XX | хх |

Table 1107 Incidence rate, number and frequency of Local AE by SAE

<sup>\*</sup>Same as Table 1102

<sup>\*</sup>Same as Table 1102

<sup>\*</sup>Same as Table 1102

<sup>\*</sup>Same as Table 1106

#### \*Same as Table 1106

Table 1109 Incidence rate, number and frequency of Local AE by Relationship \*Same as Table 1106

Table 1110 Incidence rate, number and frequency of Local AE by Action taken with the Device \*Same as Table 1106

Table 1111 Incidence rate, number and frequency of Local AE by Seriousness Criteria \*Same as Table 1106

Table 1112 Incidence rate, number and frequency of Other AE by Severity

| | Severity | n | 95% C.I. of | Eroguency | Total |
|---|---|---|---|---|---|
| | Severity | (Incidence rate) | Incidence rate | Frequency | TOtal |
| | Mild | x(x.xx%) | (x.xx,x.xx) | XX | xx |
| Medifoam | Moderate | x(x.xx%) | (x.xx,x.xx) | XX | xx |
| Wicalioalli | Severe | x(x.xx%) | (x.xx,x.xx) | XX | xx |
| | Total | x(x.xx%) | (x.xx,x.xx) | XX | xx |
| | Mild | x(x.xx%) | (x.xx,x.xx) | XX | xx |
| Betafoam | Moderate | x(x.xx%) | (x.xx,x.xx) | XX | xx |
| Betaloani | Severe | x(x.xx%) | (x.xx,x.xx) | XX | xx |
| | Total | x(x.xx%) | (x.xx,x.xx) | XX | xx |

Table 1113 Incidence rate, number and frequency of Other AE by SAE

Table 1114 Incidence rate, number and frequency of Other AE by Outcome

Table 1115 Incidence rate, number and frequency of Other AE by Relationship

Table 1116 Incidence rate, number and frequency of Other AE by Action taken with the Device \*Same as Table 1112

Table 1117 Incidence rate, number and frequency of Other AE by Seriousness Criteria

<sup>\*</sup>Same as Table 1112

<sup>\*</sup>Same as Table 1112

<sup>\*</sup>Same as Table 1112

<sup>\*</sup>Same as Table 1112